CLINICAL TRIAL: NCT05194462
Title: Home Biofeedback or Pelvic Floor Physical Therapy for Postpartum Urinary Incontinence.: A Noninferiority Randomized Controlled Trial
Brief Title: Home Biofeedback or Pelvic Floor Physical Therapy for Postpartum Urinary Incontinence.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low accrual
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jessica Sassani, Physician, Division of Urogynecology, Department of Obstetrics & Gynecology, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: POUT/IRB00297309
Record Dates: First submitted 2021-09-19; First posted 2022-01-18 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-04

CONDITIONS: Urinary Incontinence; Pelvic Floor Disorders
MeSH Terms: conditions — Urinary Incontinence; Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Pelvic Floor Physical Therapy (PFPT) (Active Comparator): 6 sessions of PFPT over a 12 week period with planned home exercises as per physical therapist's recommendation.
  Interventions: Other: Pelvic Floor Physical Therapy
- Biofeedback device (Active Comparator): Pericoach® by Analytica is a vaginal device with recommendation for daily use during the 12 week period.
  Interventions: Device: Pericoach® by Analytica

INTERVENTIONS:
Device: Pericoach® by Analytica — This intervention will assess urinary incontinence-related quality of life in postpartum women with self-reported urinary incontinence who are randomized to a program of home biofeedback .
  Arms: Biofeedback device
Other: Pelvic Floor Physical Therapy — This intervention will assess urinary incontinence-related quality of life in postpartum women with self-reported urinary incontinence who are randomized to a program of PFPT.
  Arms: Pelvic Floor Physical Therapy (PFPT)

SUMMARY:
Pelvic floor dysfunction is commonly seen in the postpartum women with symptoms including urinary urgency and frequency, urinary incontinence and fecal incontinence. Pelvic floor physical therapy (PFPT) and home biofeedback devices have been shown to improve pelvic floor symptoms in postpartum and non-postpartum populations, respectively. This randomized noninferiority clinical trial will assess urinary incontinence-related quality of life in postpartum women with self-reported urinary incontinence who are randomized to a program of home biofeedback or pelvic floor physical therapy.

DETAILED DESCRIPTION:
The objective of this proposal is to determine if home biofeedback devices are noninferior to pelvic floor physical therapy for the treatment of postpartum urinary incontinence through a randomized noninferiority clinical trial. The hypothesis is that both interventions will improve incontinence-related quality of life and that home biofeedback will be noninferior to PFPT. Two specific aims will be investigated: 1) Determine the impact of both interventions on urinary incontinence-related quality of life measured by the change in score at 3-months on the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF); 2) Determine patient impression of symptoms improvement (measured by the change in score at 3-months and 1-year on the Patient Global Impression of Improvement scale or PGI-I), overall pelvic floor symptoms (measured by the change in score at 3-months and 1-year on the Pelvic Floor Distress Inventory of PFDI) and changes in sexual function (measured by a change in score at 3-months and 1-year in the Female Sexual Function Index or FSFI). An additional exploratory aim will be to observe the change in pelvic floor symptoms in the postpartum period at 3-months and 1-year among a cohort of women who elect for the standard of care without PFPT or biofeedback.

ELIGIBILITY:
Inclusion Criteria:

* following a vaginal delivery (primiparous or multiparous, spontaneous, forceps, or vacuum assisted)
* willingness to participate in PFPT or home biofeedback exercises
* access to a smartphone with Bluetooth capabilities
* positive screen for urinary incontinence between 4 and 8 weeks postpartum defined as patient report of any urinary leakage within the prior two weeks

Exclusion Criteria:

* multiple births or deliver at ≤34 weeks
* previous urinary incontinence or pelvic organ prolapse surgery
* self-identified pre-pregnancy pelvic floor disorder such as urinary incontinence
* fecal incontinence or chronic pelvic pain or if they have a history of prior PFPT

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women age 18 of greater following a vaginal delivery.
Enrollment: 3 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-08 (Actual)

PRIMARY OUTCOMES:
Determine the impact of both interventions on urinary incontinence-related quality of life using validated questionnaire | 3 months
  Measured by the change in score on the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) between baseline and 3 months; scored between 0 and 21 with higher score meaning larger symptom burden

SECONDARY OUTCOMES:
Determine the impact of both interventions on urinary incontinence-related quality of life using validated questionnaire | 12 months
  Measured by the change in score on the International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) between baseline and 12 months; scored between 0 and 21 with higher score meaning larger symptom burden
Determine overall pelvic floor symptoms measured by validated questionnaire | 3 months
  Measured by change in score on the Pelvic Floor Distress Inventory (PFD-I) between baseline and 3 months; scored between 0 and 300 with higher score indicating greater symptom burden
Determine overall pelvic floor symptoms measured by validated questionnaire | 12 months
  Measured by change in score on the Pelvic Floor Distress Inventory (PFD-I) between baseline and 12 months; scored between 0 and 300 with higher score indicating greater symptom burden
Determine changes in sexual function following intervention measured by validated questionnaire | 3 months
  Measured by change in score on the Female Sexual Function Index (FSFI) between baseline and 3 months; scored between 2 and 36 with a lower score indicating more sexual dysfunction
Determine changes in sexual function following intervention measured by validated questionnaire | 12 months
  Measured by change in score on the Female Sexual Function Index (FSFI) between baseline and 12 months; scored between 2 and 36 with a lower score indicating more sexual dysfunction
Determine the patient impression of symptom improvement using validated questionnaire | 3 months
  Measured by the change in score on the Patient Global Impression of Improvement (PGI-I) between baseline and 3 months; scored between 1 and 7 with higher scoring meaning worsening symptoms
Determine the patient impression of symptom improvement using validated questionnaire | 12 months
  Measured by the change in score on the Patient Global Impression of Improvement (PGI-I) between baseline and 12 months; scored between 1 and 7 with higher scoring meaning worsening symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Sassani, MD, Principal Investigator — Allegheny Health Network
Locations (3):
- United States (3):
  - AHN Forbes Hospital, Monroeville, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - AHN Wexford Hospital, Wexford, Pennsylvania

IPD SHARING:
Plan to Share IPD: No
Results will be published; patient identifiers will not be used in the research publications.